CLINICAL TRIAL: NCT06215105
Title: Complex Aneurysm Registry - Real-World Evidence Data Collection Intracranial Aneurysm Treatment Devices
Acronym: CAR
Status: Enrolling by invitation | Type: Observational
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CL11025
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Aneurysm Cerebral
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Intracranial Aneurysm Devices — Intracranial Aneurysm occlusion

SUMMARY:
To collect real-world evidence allowing assessment of functional, imaging, and safety outcomes of commercially available MicroVention devices used for the endovascular treatment of intracranial aneurysms (IA) at the direction of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have a single ruptured or unruptured IA for which endovascular treatment has been determined appropriate.
2. Patient's IA will be treated using a commercially available MicroVention implant device as the primary treatment device and the decision to use this device has been made by the treating physician outside the context of the CAR study and prior to enrollment.

   Note: For the purposes of this protocol, ancillary/accessory devices such as balloon catheters and other access devices are not considered primary treatment devices.
3. Patient or patient 's legally authorized representative (LAR) has provided written informed consent prior to treatment or no later than 48 hours post procedure for emergent treatment of a ruptured aneurysm.
4. Patient must be considered by the treating physician to be available for and able to complete study follow-up visits.

Exclusion Criteria:

1. Target aneurysm has been previously treated via surgical or endovascular means.
2. Patient is enrolled in another device or drug study in which participation could confound study results.
3. Patient has a life expectancy of less than 1 year due to other illness or condition (in addition to an intracranial aneurysm).
4. Patient has been previously enrolled into this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ruptured or unruptured intracranial aneurysms who will be treated endovascularly with commercially available MicroVention devices at the direction of the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2029-01-08 (Estimated); Study Completion 2029-01-08 (Estimated)

PRIMARY OUTCOMES:
RROC | 1 year
  Angiographic aneurysm occlusion (RROC) at 1 year
RROC | 1 year
  Angiographic aneurysm occlusion (RROC) at 1 year without rebleed (ruptured aneurysms only)
RROC | 1 year
  Angiographic aneurysm occlusion (RROC) at 1 year without rebleed (ruptured aneurysms only) or retreatment for residual aneurysm

CONTACTS AND LOCATIONS:
Overall Officials: TBD TBD, Principal Investigator
Locations (5):
- United States (5):
  - Memorial Healthcare System, Hollywood, Florida
  - Orlando Health, Orlando, Florida
  - University of Iowa, Iowa City, Iowa
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Albany Medical Center, Albany, New York